CLINICAL TRIAL: NCT06123026
Title: Pharmacological Inhibition of Lactation After 16 to 20 Week Abortion: a Randomized Controlled Trial
Brief Title: Pharmacological Inhibition of Lactation After 16 to 20 Week Abortion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00218555
Record Dates: First submitted 2023-10-28; First posted 2023-11-08 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Lactation Suppressed; Second Trimester Abortion
MeSH Terms: interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabergoline (Experimental): 1mg oral cabergoline administered once after patient's procedure
  Interventions: Drug: Cabergoline
- Placebo (Placebo Comparator): 1 tablet encapsulated placebo by Investigational Drug Pharmacy administered once after patient's procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cabergoline — 1mg oral cabergoline given to participants once
  Arms: Cabergoline
Drug: Placebo — 1 encapsulated placebo tablet given to participants after procedure
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare breast symptoms (lactation, engorgement, etc) of individuals who undergo a procedure for second trimester of pregnancy loss between 16 weeks and 20 weeks gestational age. The participants will be randomly placed in two groups, one with a placebo tablet and one with medication called "cabergoline" which are taken immediately after their procedure. Researchers will compare groups to see if there are any significant differences in breast symptoms.

ELIGIBILITY:
Inclusion Criteria:

* pregnant individuals seeking termination of pregnancy after 16w0d gestation and up to 19w6d gestation. this includes management of intrauterine demises
* ages 18 to 50
* con provide informed consent in English

Exclusion Criteria:

* Age under 18 or above 50
* gestational ages before 16 weeks 0 days or after 20 weeks 0 days
* unable to provide written consent in English
* hypertensive disorder
* uncontrolled hypertension or known hypersensitivity to ergot derivatives
* History of cardiac valvular disorders
* history of pulmonary fibrosis
* documented bipolar schizophrenia
* documented allergy to medication, including lactose intolerance (placebo pill involves lactose)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
breast symptoms | 3 days post procedure and two weeks post procedure
  Using the bristol breast inventory to assess breast symptoms (engorgement, lactation, etc).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No